CLINICAL TRIAL: NCT03099551
Title: Randomized Trial to Evaluate the Efficacy of Two Different Toothbrushes on Plaque Control
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Faculty Sao Leopoldo Mandic Campinas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1.672.795
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Plaque; Gingivitis
Keywords: Plaque; oral hygiene; gingivitis; sonic toothbrush; manual toothbrush
MeSH Terms: conditions — Plaque, Amyloid; Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Toothbrush users (Active Comparator): Group using manual toothbrush Curaprox 5460 Ultra Soft
  Interventions: Device: Group using manual toothbrush Curaprox 5460 Ultra Soft
- Sonic Toothbrush users (Active Comparator): Group using sonic toothbrush Edel White
  Interventions: Device: Group using sonic toothbrush Edel White

INTERVENTIONS:
Device: Group using manual toothbrush Curaprox 5460 Ultra Soft — Manual toothbrush usage with Bass technique twice a day during 2 minutes
  Arms: Manual Toothbrush users
Device: Group using sonic toothbrush Edel White — Sonic toothbrush usage twice a day during 2 minutes
  Arms: Sonic Toothbrush users

SUMMARY:
The aim of the present study was to evaluate the efficacy of two different toothbrushes (manual and sonic) on plaque control

DETAILED DESCRIPTION:
A parallel randomized clinical trial, examiner-blind, was conducted involving 56 patients with ages from 15 to 20, all students of CAMP (Centro de Formação e Integração Social), in the city of São Bernardo do Campo, state of São Paulo, Brazil. Randomization: the subjects were randomly allocated to two different groups (A for the manual toothbrush and B for the sonic toothbrush) by removing from an urn a paper with their respective group. Silness & Löe Gingival Index, the Turesky Modification of the Quigley Hein Plaque Index and the Community Periodontal Index were evaluated at baseline and after 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects had to be in generally good health, and possessing a minimum of 20 permanent natural teeth, excluding third molars.

Exclusion Criteria:

* Subjects were excluded if they had fixed orthodontic appliances, advanced periodontal disease, limited manual dexterity, active caries, medical conditions limiting their salivary function or immunological condition, and if they were smokers.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Silness & Löe Gingival Index | 6 months
  0 = Normal gingiva; 1 = Mild inflammation - slight change in colour, slight oedema. No bleeding on probing; 2 = Moderate inflammation - redness, oedema and glazing; bleeding on probing; 3 = Severe inflammation - marked redness and oedema. Ulceration. Tendency to spontaneous bleeding
Turesky Modification of the Quigley Hein Plaque Index | 6 months
  0 = No plaque; 1 = Separate flecks of plaque at the cervical margin of the tooth; 2 = A thin continuous band of plaque (up to one mm) at the cervical margin of the tooth; 3 = A band of plaque wider than one mm but covering less than one third of the crown of the tooth; 4 = Plaque covering at least one-third but less than two-thirds of the crown of the tooth; 5 = Plaque covering two-thirds or more of the crown of the tooth
Community periodontal index | 6 months
  0 = No periodontal disease; 1 = Bleeding on probing; 2 = Calculus with plaque seen or felt by probing.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aass AM, Gjermo P. Comparison of oral hygiene efficacy of one manual and two electric toothbrushes. Acta Odontol Scand. 2000 Aug;58(4):166-70. doi: 10.1080/000163500429163. PMID 11045370
- [Background] Araujo AC, Gusmao ES, Batista JE, Cimoes R. Impact of periodontal disease on quality of life. Quintessence Int. 2010 Jun;41(6):e111-8. PMID 20490384
- [Background] Ayad F, Petrone DM, Wachs GN, Mateo LR, Chaknis P, Panagakos F. Comparative efficacy of a specially engineered sonic powered toothbrush with unique sensing and control technologies to two commercially available power toothbrushes on established plaque and gingivitis. J Clin Dent. 2012;23 Spec No A:A5-10. PMID 23448082
- [Background] Barros VA, Costa SM, Zanin L, Florio FM. Evaluation of an educational activity in the oral health of students. Int J Dent Hyg. 2017 Feb;15(1):23-29. doi: 10.1111/idh.12152. Epub 2015 Jun 5. PMID 26053214
- [Background] BASS CC. The optimum characteristics of toothbrushes for personal oral hygiene. Dent Items Interest. 1948 Jul;70(7):697-718. No abstract available. PMID 18871313
- [Background] Borges Tde F, Regalo SC, Taba M Jr, Siessere S, Mestriner W Jr, Semprini M. Changes in masticatory performance and quality of life in individuals with chronic periodontitis. J Periodontol. 2013 Mar;84(3):325-31. doi: 10.1902/jop.2012.120069. Epub 2012 May 1. PMID 22548588
- [Background] Castro CO, Katiane SO, Carvalho RB, Garbin CAS, Bueno RN. Education and prevention programs for oral health in schools: a critical analysis of national publications. OdontolClín-Cient 2012 Jan-Mar; 11(1): 35-9.
- [Background] Baccareli JC, Ribeiro MC. Sensibilidade dos Lactobacillus a anti-sépticos bucais. Rev Cienc Med, Campinas 2000; 9(3):99-104.
- [Background] Chalub LLF, Péret ACA. Desempenho do Índice Periodontal Comunitário (CPI) na determinação da condição periodontal: enfoque no exame parcial. Revista do Arquivo Brasileiro de Odontologia. 2010;6(3):155-62.
- [Background] Cifcibasi E, Koyuncuoglu CZ, Baser U, Bozacioglu B, Kasali K, Cintan S. Comparison of manual toothbrushes with different bristle designs in terms of cleaning efficacy and potential role on gingival recession. Eur J Dent. 2014 Jul;8(3):395-401. doi: 10.4103/1305-7456.137655. PMID 25202222
- [Background] Erbe C, Klukowska M, Tsaknaki I, Timm H, Grender J, Wehrbein H. Efficacy of 3 toothbrush treatments on plaque removal in orthodontic patients assessed with digital plaque imaging: a randomized controlled trial. Am J Orthod Dentofacial Orthop. 2013 Jun;143(6):760-6. doi: 10.1016/j.ajodo.2013.03.008. PMID 23726325
- [Background] Fjeld KG, Mowe M, Eide H, Willumsen T. Effect of electric toothbrush on residents' oral hygiene: a randomized clinical trial in nursing homes. Eur J Oral Sci. 2014 Apr;122(2):142-8. doi: 10.1111/eos.12113. Epub 2014 Jan 20. PMID 24438077
- [Background] Goyal CR, Qaqish J, He T, Grender J, Walters P, Biesbrock AR. A randomized 12-week study to compare the gingivitis and plaque reduction benefits of a rotation-oscillation power toothbrush and a sonic power toothbrush. J Clin Dent. 2009;20(3):93-8. PMID 19711610
- [Background] Goyal CR, Klukowska M, Grender JM, Cunningham P, Qaqish J. Evaluation of a new multi-directional power toothbrush versus a marketed sonic toothbrush on plaque and gingivitis efficacy. Am J Dent. 2012 Sep;25 Spec No A(A):21A-26A. PMID 23248895
- [Background] Grender J, Williams K, Walters P, Klukowska M, Reick H. Plaque removal efficacy of oscillating-rotating power toothbrushes: review of six comparative clinical trials. Am J Dent. 2013 Apr;26(2):68-74. PMID 24073528
- [Background] Hashim R, Williams S, Thomson WM. Oral hygiene and dental caries in 5- to 6-year-old children in Ajman, United Arab Emirates. Int J Dent Hyg. 2013 Aug;11(3):208-15. doi: 10.1111/idh.12011. Epub 2012 Dec 6. PMID 23216907
- [Background] Jin LJ, Armitage GC, Klinge B, Lang NP, Tonetti M, Williams RC. Global oral health inequalities: task group--periodontal disease. Adv Dent Res. 2011 May;23(2):221-6. doi: 10.1177/0022034511402080. PMID 21490234
- [Background] Kinane DF, Berglundh T, Lindhe J. Patogênese da Pariodontite. In: Lindhe J, Lang N. P, Karring T. Tratado de Periodontia Clínica e Implantologia Oral. 5a ed. Rio de Janeiro: Guanabara Koogan; 2010. P.271-91.
- [Background] Klukowska M, Grender JM, Timm H. A single-brushing study to compare plaque removal efficacy of a new power brush to an ADA reference manual toothbrush. Am J Dent. 2012 Sep;25 Spec No A(A):10A-13A. PMID 23248893
- [Background] Klukowska M, Grender JM, Conde E, Goyal CR. A 12-week clinical comparison of an oscillating-rotating power brush versus a marketed sonic brush with self-adjusting technology in reducing plaque and gingivitis. J Clin Dent. 2013;24(2):55-61. PMID 24282870
- [Background] Klukowska M, Grender JM, Conde E, Ccahuana-Vasquez RA, Goyal CR. A randomized 12-week clinical comparison of an oscillating-rotating toothbrush to a new sonic brush in the reduction of gingivitis and plaque. J Clin Dent. 2014;25(2):26-31. PMID 25122979
- [Background] Klukowska M, Grender JM, Conde E, Ccahuana-Vasquez RA, Ram Goyal C. A randomized clinical trial evaluating gingivitis and plaque reduction of an oscillating-rotating power brush with a new brush head with angled bristles versus a marketed sonic brush with self-adjusting technology. Am J Dent. 2014 Aug;27(4):179-84. PMID 25831599
- [Background] Klukowska M, Grender JM, Conde E, Goyal CR, Qaqish J. A six-week clinical evaluation of the plaque and gingivitis efficacy of an oscillating-rotating power toothbrush with a novel brush head utilizing angled CrissCross bristles versus a sonic toothbrush. J Clin Dent. 2014;25(2):6-12. PMID 25122976
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Lopes MWF, Gusmão ES, Alves RV, Cimões R. The Impacto f Chronic Periodontitis on Quality of Life in Brazilian Subjects. Acta Stomatol Croat. 2009 June;43(2):89-98.
- [Background] Marinho BVS, Araújo ACS. Uso dos enxaguatórios bucais sobre a gengivite e biofilme dental. International Journal of Dentistry 2007; 6(4):124-31.
- [Background] Marini I, Bortolotti F, Parenti SI, Gatto MR, Bonetti GA. Combined effects of repeated oral hygiene motivation and type of toothbrush on orthodontic patients: a blind randomized clinical trial. Angle Orthod. 2014 Sep;84(5):896-901. doi: 10.2319/112113-856.1. Epub 2014 Mar 18. PMID 24641783
- [Background] Meusel DR, Ramacciato JC, Motta RH, Brito Junior RB, Florio FM. Impact of the severity of chronic periodontal disease on quality of life. J Oral Sci. 2015 Jun;57(2):87-94. doi: 10.2334/josnusd.57.87. PMID 26062856
- [Background] Moritis K, Jenkins W, Hefti A, Schmitt P, McGrady M. A randomized, parallel design study to evaluate the effects of a Sonicare and a manual toothbrush on plaque and gingivitis. J Clin Dent. 2008;19(2):64-8. PMID 18763689
- [Background] Nathoo S, Mankodi S, Mateo LR, Chaknis P, Panagakos F. A clinical study comparing the supragingival plaque and gingivitis efficacy of a specially engineered sonic powered toothbrush with unique sensing and control technologies to a commercially available manual flat-trim toothbrush. J Clin Dent. 2012;23 Spec No A:A11-6. PMID 23448083
- [Background] Nightingale KJ, Chinta SK, Agarwal P, Nemelivsky M, Frisina AC, Cao Z, Norman RG, Fisch GS, Corby P. Toothbrush efficacy for plaque removal. Int J Dent Hyg. 2014 Nov;12(4):251-6. doi: 10.1111/idh.12081. Epub 2014 Apr 17. PMID 24738786
- [Background] Papapanou PN, Lindhe J. Epidemiologia das doenças periodontais. In: Lindhe J, Lang NP, Karring T. Tratado de Periodontia Clínica e Implantologia Oral. 5a ed. Rio de Janeiro: Guanabara Koogan; 2010. p.123-70.
- [Background] Parizi MT, Mohammadi TM, Afshar SK, Hajizamani A, Tayebi M. Efficacy of an electric toothbrush on plaque control compared to two manual toothbrushes. Int Dent J. 2011 Jun;61(3):131-5. doi: 10.1111/j.1875-595X.2011.00029.x. PMID 21692783
- [Background] Pedrazzi V; Souza, SLS, Oliveira RR; Cimões R; Gusmão ES. Métodos mecânicos para o controle do biofilme dentário supragengival. Periodontia;19(3):26-33, 2009.
- [Background] Peng Y, Wu R, Qu W, Wu W, Chen J, Fang J, Chen Y, Farella M, Mei L. Effect of visual method vs plaque disclosure in enhancing oral hygiene in adolescents and young adults: a single-blind randomized controlled trial. Am J Orthod Dentofacial Orthop. 2014 Mar;145(3):280-6. doi: 10.1016/j.ajodo.2013.10.021. PMID 24582019
- [Background] Pizzo G, Licata ME, Pizzo I, D'Angelo M. Plaque removal efficacy of power and manual toothbrushes: a comparative study. Clin Oral Investig. 2010 Aug;14(4):375-81. doi: 10.1007/s00784-009-0303-3. Epub 2009 Jun 23. PMID 19548011
- [Background] QUIGLEY GA, HEIN JW. Comparative cleansing efficiency of manual and power brushing. J Am Dent Assoc. 1962 Jul;65:26-9. doi: 10.14219/jada.archive.1962.0184. No abstract available. PMID 14489483
- [Background] Re D, Augusti G, Battaglia D, Gianni AB, Augusti D. Is a new sonic toothbrush more effective in plaque removal than a manual toothbrush? Eur J Paediatr Dent. 2015 Mar;16(1):13-8. PMID 25793947
- [Background] Rufasto Goche K, Saavedra Alvarado B. Aplicación de un programa educativo en salud oral en adolescentes de una institución educativa peruana. Rev Estomatol Herediana 2012 abr-jun; ;22(2):82-90.
- [Background] Soares D, Andrade A, Pinto AR, Seabra M, Macho V. Doenças da gengiva e periodonto em crianças e adolescentes. Acta Pediatr Port 2009 40(1):23-29.
- [Background] Saba-Chujfi E, Silva ECQ, Sarian R. Avaliação dos métodos de motivação/educação em higiene bucal. RGO. 1992; 40:87-90.
- [Background] Schmickler J, Wurbs S, Wurbs S, Lange K, Rinke S, Hornecker E, Mausberg RF, Ziebolz D. Influence of the utilization time of different manual toothbrushes on oral hygiene assessed during a 6-month observation period: a randomized clinical trial. J Periodontol. 2014 Aug;85(8):1050-8. doi: 10.1902/jop.2013.130442. Epub 2013 Dec 12. PMID 24329045
- [Background] Swierkot K, Brusius M, Leismann D, Nonnenmacher C, Nusing R, Lubbe D, Schade-Brittinger C, Mengel R. Manual versus sonic-powered toothbrushing for plaque reduction in patients with dental implants: an explanatory randomised controlled trial. Eur J Oral Implantol. 2013 Summer;6(2):133-44. PMID 23926585
- [Background] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376
- [Background] Williams K, Rapley K, Haun J, Walters P, Grender J, He T, Biesbrock AR. Benefit of the power component of sonic and rotation-oscillation modes of action for plaque removal using power toothbrushes. Am J Dent. 2010 Apr;23(2):60-4. PMID 20608293
- [Background] World Health Organization. Health Promotion: A Discussion Document on the Concept and Principles. Copenhagen: WHO Regional Office for Europe, 1984
- [Background] World Health Organization. Oral health surveys: basic methods. 5th Ed. Geneva: World Health Organization; 2013.
- See also: Brazil. Ministry of Health. Healthcare Department/Health Inspection Office. Department of Basic Healthcare. General Management of Oral Health. SBBrasil: principal results. Brasília: Ministry of Health; 2010. — http://dab.saude.gov.br/CNSB/sbbrasil/arquivos/projeto_sb2010_relatorio_final.pdf